CLINICAL TRIAL: NCT06577948
Title: Spectacle Lenses Utilising P.A.U.S.E.® Technology for Slowing Down Myopia Progression in Vietnamese Children: a Prospective, Masked, Controlled, Randomised, Clinical Trial
Brief Title: The P.A.U.S.E.® Spectacle Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: nthalmic Pty Ltd (Network)
Collaborators: Brighten Optix Corporation (Unknown)
Responsible Party: Principal Investigator, Daniel Tilia, MOptom, PhD, Principal Research Optometrist, nthalmic Pty Ltd
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: nthal2024-01
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Myopia
Keywords: axial length
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Investigators, participants, and parents/legal guardians will be masked to the identity of the study product worn by each participant. All spectacle lenses will be fitted into the chosen spectacle frame. P.A.U.S.E.® optical elements may be visible under certain lighting conditions, and therefore, it may not be possible to completely mask test spectacle lenses from control spectacle lenses. However, complete masking is possible between test spectacle lenses. Regardless, investigators who perform crucial measurements (axial length and autorefraction) should not view a participant's study product to further minimise the chance of de masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Assigned Intervention 1 (Active Comparator): Single vision spectacle lens
  Interventions: Device: Single vision spectacle lens
- Assigned Intervention 2 (Experimental): P.A.U.S.E. spectacle lens 1
  Interventions: Device: P.A.U.S.E. spectacle lens 1
- Assigned Intervention 3 (Experimental): P.A.U.S.E. spectacle lens 2
  Interventions: Device: P.A.U.S.E. spectacle lens 2

INTERVENTIONS:
Device: Single vision spectacle lens — Standard single vision spectacle lens
  Arms: Assigned Intervention 1
Device: P.A.U.S.E. spectacle lens 1 — P.A.U.S.E. spectacle lens 1
  Arms: Assigned Intervention 2
Device: P.A.U.S.E. spectacle lens 2 — P.A.U.S.E. spectacle lens 2
  Arms: Assigned Intervention 3

SUMMARY:
The goal of this clinical trial is to learn if spectacle lenses using Phase Alteration Utilising Sub Elements (P.A.U.S.E.®) technology works to slow down the rate of myopia progression compared to single vision spectacle lenses in myopic children. The main questions it aims to answer are:

Do spectacle lenses using P.A.U.S.E.® technology slow down the rate of axial length growth? Do spectacle lenses using P.A.U.S.E.® technology slow down the rate of increase in myopic refractive error?

Researchers will compare spectacle lenses using P.A.U.S.E.® technology to a single vision spectacle lens.

Participants will:

Be randomly allocated to wear either spectacle lenses using P.A.U.S.E.® technology or single vision spectacle lenses.

Visit the clinic on five occasions over a 12 month period.

DETAILED DESCRIPTION:
The aim of this clinical trial is to compare the rate of myopia progression as measured by change from the Dispensing visit (up to 26 days from Baseline), in axial length and the change from Baseline in the spherical equivalent cycloplegic autorefraction between two spectacle lens designs using P.A.U.S.E.® technology (tests) and single vision spectacle lenses ( control). Myopic children (6-14 years of age) will be randomly allocated to wear either test 1, test 2, or control.

The overall trial duration, including follow-up period, is expected to be approximately 18 months. Each participant's duration is expected to be approximately 12 months.

The visits are Baseline, Dispensing, 1 month, 6 months, and 12 months.

All procedures performed at these visits are standard, non invasive clinical tests.

ELIGIBILITY:
Inclusion Criteria:

* Be between 6-14 years inclusive at time of enrolment.
* Have:

  * Read the Informed Assent.
  * Been explained the Informed Assent.
  * Indicated an understanding of the Informed Assent.
  * Signed the Informed Assent.
* Have their parent / legal guardian:

  * Read the Informed Consent.
  * Been explained the Informed Consent.
  * Indicated an understanding of the Informed Consent.
  * Signed the Informed Consent.
* Along with their parent / legal guardian, be capable of comprehending the nature of the study, and be willing and able to adhere to study requirements.
* Along with their parent / legal guardian, agree to maintain the visit and prescribed wearing schedule.
* Agree to wear allocated spectacles for a minimum of 5 days per week, at least 6 hours per day for the duration of the study and to inform the investigator if their schedule is interrupted.
* Be in good general health, based on the parent's / legal guardian's knowledge.
* Have best-corrected high contrast visual acuity based on manifest refraction of 0.10 logMAR (Snellen: 20/25, 6/7.6; Decimal: 0.8) or better in each eye.
* Meet the following criteria determined by cycloplegic autorefraction at Baseline:

  o-5.00 D ≤ spherical equivalent ≤ -0.75 D and sphere component ≤ -0.50 DS. o-1.50 DC ≤ astigmatic component ≤ 0 DC. o|Spherical equivalent anisometropia| ≤ 1.00 D.

Exclusion Criteria:

* Participant is currently an active participant in another study or was active participant in another study within 30 days prior to this study.
* Current or prior use of interventions intended for myopia control, including but not limited to:

  * Optical devices:

    * Bifocal / multifocal spectacles.
    * Bifocal / multifocal contact lenses.
    * Orthokeratology.
  * Pharmacological agents:

    * Atropine with a concentration > 0.01%.
    * Participants who have previously used 0.01% atropine are eligible for this study provided they agree not to use 0.01% atropine for at least 30 days before baseline and at any time during the study.
    * Pirenzepine.
* Participant born earlier than 30 weeks or weighed < 1500 g at birth.

  o A verbal report from the participant's parent / legal guardian is sufficient.
* Habitual use of a systemic or topical medication that may alter normal ocular findings / is known to affect a participant's ocular health / physiology either in an adverse or beneficial manner at enrolment and / or during the clinical trial.
* A known allergy to sodium fluorescein, benoxinate, proparacaine, tropicamide, or cyclopentolate.
* Strabismus as determined by cover test at distance (≥ 3 m) or near (40 cm) while wearing distance correction under non-cycloplegic conditions.
* Known ocular or systemic disease, such as but not limited to:

  * Diabetes.
  * Graves' disease.
  * Glaucoma.
  * Uveitis.
  * Scleritis.
  * Auto-immune diseases such as ankylosing spondylitis, multiple sclerosis, Sjogren's syndrome, and systemic lupus erythematosus.
* Any ocular, systemic, or neuro-developmental conditions that could influence refractive development, such as but not limited to:

  * Persistent pupillary membrane.
  * Vitreous haemorrhage.
  * Cataract.
  * Central corneal scarring.
  * Eyelid haemangiomas.
  * Marfan's syndrome.
  * Down's syndrome.
  * Ehler's-Danlos syndrome.
  * Stickler's syndrome.
  * Ocular albinism.
  * Retinopathy of prematurity.
* Keratoconus or irregular cornea.
* The investigator may, at their discretion, exclude anyone who they believe may not be able to fulfil the clinical trial requirements or it is believed to be in the participant's best interests.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 250 (Estimated)
Dates: Start 2024-09-14 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Axial Length | Dispensing Visit (up to 26 days from Baseline), then 1 month, 6 months, and 12 months after Dispensing Visit
  Difference in change from dispensing in axial length between each test and control.

SECONDARY OUTCOMES:
Cycloplegic spherical equivalent autorefraction | Baseline, then 6 months, and 12 months after Dispensing Visit (up to 26 days from Baseline).
  Difference in change from Baseline in cycloplegic spherical equivalent autorefraction between each test and control.
Visual performance as measured by high contrast visual acuity at 6 m | Dispensing Visit (up to 26 days from Baseline), then 1 month, 6 months, and 12 months after Dispensing Visit
  Difference in visual acuity between each test and control.
Visual performance as measured by a non validated questionnaire based on a 1-10 | 1 month, 6 months, and 12 months after Dispensing Visit (up to 26 days from Baseline).
  Difference in subjective visual performance between each test and control.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Tilia, MOptom, PhD, Principal Investigator — nthalmic Pty Lyd
Locations (1):
- Hai Yen Eye Care, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available to other researchers.